CLINICAL TRIAL: NCT07390279
Title: Efficacy of Transcutaneous Pulsed Radiofrequency in Postherpetic Neuralgia
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Salim Taner Gözükızıl, Pain specialist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: Postherpetic Neuralgia
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Postherpetic Neuralgia; Chronic Pain; Neuropathy
Keywords: postherpetic neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transcutaneous Pulsed Radiofrequency — The TCPRF procedure will be performed by the same algology specialist. Patients will be monitored according to standard protocols, including noninvasive blood pressure, pulse oximetry, and electrocardiography. The procedure will be conducted in the supine position. For TCPRF, 45 × 98 mm transcutaneous electrodes (Equip, FIAB SPA, Via P. Costoli, Italy) will be used. Electrodes will be placed over the most painful area along the affected dermatome. TCPRF will be delivered at 80 volts, 2 Hz, and 20 ms pulse width for a duration of 8 minutes. The procedure will be repeated three times at one-week intervals.

SUMMARY:
Postherpetic neuralgia (PHN) is a chronic pain syndrome that may be resistant to treatment and can lead to physical and social disability as well as psychological disturbances, persisting for years in some patients. Varicella zoster virus remains latent in the sensory neurons of individuals who have previously had chickenpox. Reactivation of the latent virus results in herpes zoster. Herpes zoster typically begins with dermatomal pain, followed within a few days by the development of characteristic dermatomal skin rashes. These cutaneous lesions usually resolve within 2-4 weeks; however, pain may persist even after the rash has healed.

There is variability in the literature regarding the definition of PHN. The development of PHN is associated with increased central neuronal sensitization, reduced inhibitory neuronal function, inflammation and nerve injury in the peripheral nervous system, and abnormal neural transmission following nerve damage. PHN is the most common complication of herpes zoster and occurs in approximately 9-19% of affected patients. Its incidence increases with age, occurring in about 2% of patients under 50 years of age, approximately 20% of those over 50 years, and nearly 35% of patients over 80 years of age.

Various treatment options are available for the management of PHN-related pain, including pharmacological and interventional approaches. Systemic agents include tricyclic antidepressants, calcium channel alpha-2-delta ligands, serotonin-norepinephrine reuptake inhibitors, and opioids, while topical treatments include lidocaine and capsaicin. Interventional treatment options for PHN include epidural and intrathecal injections, sympathetic nerve blocks, erector spinae plane block, subcutaneous injections, and spinal cord stimulation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the analgesic efficacy of Transcutaneous Pulsed Radiofrequency (TCPRF), a non-invasive neuromodulation technique, in adult patients diagnosed with postherpetic neuralgia (PHN) who are refractory to conventional treatments. The study aims to prospectively assess the pain-reducing effect of TCPRF applied to the affected dermatomal area by comparing pain intensity, measured using Visual Analog Scale (VAS) scores, at 1 and 3 months after the procedure with baseline values.

The secondary objectives of the study are to comprehensively evaluate the effects of TCPRF treatment on both the sensory (e.g., throbbing, stabbing) and affective (e.g., tiring, fearful) dimensions of pain using the Short-Form McGill Pain Questionnaire (SF-MPQ). In addition, changes in neuropathic pain scores assessed by the Douleur Neuropathique 4 (DN4) questionnaire and improvements in overall quality of life measured by the Short Form-12 (SF-12) will be examined. As an indicator of procedural safety, the study also aims to report any potential adverse effects or complications that may occur during or after the intervention.The study is planned to be conducted as a prospective observational study at the Algology Clinic of Cemil Taşcıoğlu City Hospital. Following the acquisition of informed consent, patients presenting to our clinic with postherpetic neuralgia will receive transcutaneous pulsed radiofrequency (TCPRF) treatment applied to the painful area. During post-treatment outpatient follow-up visits, the effects of the intervention on pain scores and quality of life will be evaluated.

As implied by its name, the procedure is performed transcutaneously via adhesive skin electrodes and does not involve any incision or invasive intervention. The planned duration of the study is six months.

In routine clinical practice, patients presenting with postherpetic neuralgia initially receive medical treatment, while interventional therapies are considered for those with insufficient or limited response to pharmacological management. These interventional options include nerve blocks, epidural injections, radiofrequency treatments, and spinal cord stimulation procedures. The TCPRF procedure performed in our clinic is part of routine clinical practice, and no additional interventional procedures will be applied to patients solely for research purposes.

Patients aged 18 years and older diagnosed with postherpetic neuralgia will be included in the study. No control group or involvement of additional medical specialties is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of postherpetic neuralgia (PHN)
* No invasive or noninvasive treatment related to PHN (e.g., capsaicin, lidocaine patches) within the past 3 months
* Provision of written informed consent

Exclusion Criteria:

* Patients with a cardiac pacemaker
* Known allergy to transcutaneous electrode pads
* Active skin infection at the pad application site
* Presence of a metallic implant in the treatment area
* Circulatory disorders or skin lesions at the treatment site
* Inability to maintain appropriate positioning
* Inability to communicate effectively
* Presence of psychosis or progressive neurological deficits
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at the Algology Department of Istanbul Cemil Taşcıoğlu City Hospital, following approval by the institutional ethics committee, and will include patients aged 18 years and older diagnosed with postherpetic neuralgia (PHN) who are scheduled to receive transcutaneous pulsed radiofrequency (TCPRF) treatment in three sessions.
  Within the scope of the study, the following data will be recorded: age, sex, body mass index (BMI), side of the procedure, history of herpes zoster vaccination (live or recombinant), family history of herpes zoster, immunosuppression status (e.g., HIV infection, malignancy, steroid use), duration of symptoms, dermatome treated with TCPRF, TCPRF-related complications and adverse effects, Visual Analog Scale (VAS) scores, neuropathic pain assessment using the Douleur Neuropathique 4 (DN4) questionnaire, and health-related quality of life assessed using the Short Form-12 (SF-12).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 months
  This scale allows for the numerical determination of the subjective intensity of pain by asking patients to rate their pain severity on a 10 cm line from 0 (no pain) to 10 (the most severe pain I have ever felt).

SECONDARY OUTCOMES:
Neuropathic Pain Questionnaire-4 | 3 months
  This is a Turkish-validated diagnostic screening test consisting of 10 items in total: 7 symptoms based on patient description and 3 clinical findings based on physical examination, which helps differentiate neuropathic pain from nociceptive pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Prof. Dr. Cemil Taşcioğlu City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No